CLINICAL TRIAL: NCT04654221
Title: Evaluation of eGFR, Determined by Cystatin C and Creatinine, and mGFR, Measured by Iohexol Clearance, in Subjects at High Risk for Acute Kidney Injury (AKI) Following Cardiac Surgery
Brief Title: Evaluation of Renal Function in Subjects Who Had Undergone Cardiac Surgery
Status: Terminated | Type: Observational
Why Stopped: Study terminated early due to program discontinuation.
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: QRK509
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Surgery
Keywords: GFR; Acute Kidney Injury; AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Male, BMI <= 24.9: Male subjects with a BMI of less than or equal to 24.9
  Interventions: Diagnostic Test: mGFR by iohexol clearance
- Female, BMI <= 24.9: Female subjects with a BMI of less than or equal to 24.9
  Interventions: Diagnostic Test: mGFR by iohexol clearance
- Male, BMI 25-29: Male subjects with a BMI of 25 to 29
  Interventions: Diagnostic Test: mGFR by iohexol clearance
- Female, BMI 25-29: Female subjects with a BMI of 25 to 29
  Interventions: Diagnostic Test: mGFR by iohexol clearance
- Male, BMI >29: Male subjects with a BMI of greater than 29
  Interventions: Diagnostic Test: mGFR by iohexol clearance
- Female, BMI >29: Female subjects with a BMI of greater than 29
  Interventions: Diagnostic Test: mGFR by iohexol clearance

INTERVENTIONS:
Diagnostic Test: mGFR by iohexol clearance — Iohexol 5mL injection (300 mg iodine/mL) will be administered to all subjects to determine mGFR by iohexol clearance

SUMMARY:
To evaluate the differences between serum cystatin C based estimated glomerular filtration rate (eGFRcys), serum creatinine based eGFR (eGFRcreat) and measured glomerular filtration rate (mGFR) in subjects at high risk for acute kidney injury (AKI) approximately 90 days following cardiac surgery

DETAILED DESCRIPTION:
This is an open label, single-visit study to evaluate the relationship between mGFR and eGFR based either on serum creatinine (eGFRcreat) or cystatin C (eGFRcys) approximately 90 days following cardiac surgery. No investigational study drug will be administered.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, age ≥ 45 years old
* At risk for AKI following cardiac surgery on the basis of at least one of the following pre-operatively assessed risk factors:

  1. Reduced renal function
  2. Diabetes with ongoing insulin treatment
  3. Albuminuria
* Have undergone non-emergent open chest cavity cardiovascular surgeries, with use of cardiopulmonary bypass (CPB), with or without hypothermic circulatory arrest

Key Exclusion Criteria:

* Emergent surgeries, including aortic dissection, and major congenital heart defects
* Past cardiac surgery off CPB
* Have a known allergy to iohexol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone non-emergent cardiac surgery and were at high risk of developing AKI, who meet all of the Inclusion and none of the Exclusion criteria, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Correlation between eGFR and mGFR | at 90 days post cardiac surgery
  The primary measure will be the comparison of the P(30) and P(10) between eGFR based on serum cystatin C (eGFRcys) and eGFR based on serum creatinine (eGFRcreat). P(30) and P(10) are defined as the percentage of subjects whose eGFR is within 30% (10%) of the iohexol-based mGFR.

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Halevy, MD, Study Director — Quark Pharmaceuticals
Locations (6):
- United States (6):
  - CB Flock Research, Mobile, Alabama
  - Valley Clinical Trials, Covina, California
  - Valley Clinical Trials, Northridge, California
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Advance Medical Research, St. Petersburg, Florida
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No